CLINICAL TRIAL: NCT06866184
Title: Regenerative Effects of Young Immortalized and Engineered MSC-Derived EVs on Aging and Senescent Brain Models
Brief Title: Regenerative Effects of Birth Material Derived Extracellular Vesicles
Acronym: ReGAIN
Status: Not yet recruiting | Type: Observational
Sponsor: University of Aberdeen (Other)
Responsible Party: Sponsor
Other Study IDs: 2-073-23; IRAS project ID: 331602 (Other: The Integrated Research Application System (IRAS), UK)
Record Dates: First submitted 2025-02-06; First posted 2025-03-10 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Caesarean Delivery
Keywords: child birth; caesarean section; healthy donor; umbilical cord; placenta

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — stem cells and extracellular vesicles obtained from birth material
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Expectant healthy females undergoing a planned Caesarean Section (full term)

SUMMARY:
Stem cells offer great hope for a wide range of disorders, including age-related brain disease such as dementia. Mesenchymal stem cells (MSCs) are special types of adult stem cells found in various tissues like the umbilical cord, placenta and bone marrow. These cells can develop into different cell types, such as bone, cartilage, muscle, and neurones. They can promote healing, regulate the immune system and repair damaged tissues. Extracellular vesicles (EVs) are tiny, bubble-like structures released by MSCs, which help communication between tissues and organs by delivering specific instructions and regenerative substances. Therefore, MSC-EVs are thought to be responsible for many of beneficial effects.

Recent evidence suggests that specific properties of EVs depend on where the MSCs come from, how old the donor was, and the environment/conditions they are in. To better understand the best source of MSC-EVs for treating age-related brain diseases, the investigators here plan to use placenta, amniotic fluid, and umbilical cord tissues of consenting mothers, who are undergoing an elective Caesarean section. Such birth tissues are rich sources of stem cells and would normally be disposed off. The investigators will here extract and analyse EVs and seek to identify the most effective ones for regenerating aged or damaged brain cells. Once the investigators identify the best source, they will seek to stabilise ("immortalize") the stem cells so that they offer a consistent source of effective MSC-EVs. Additionally, the investigators aim to modify MSCs genetically or via exposure to regenerative compounds to enhance their therapeutic properties. Promising MSC-EVs will be tested on cell culture models of brain aging and disease to validate if they can repair damage or aid recovery.

Overall, the project aims to explore sources and properties of MSC-EVs that may offer new therapeutic ways to treat brain diseases.

ELIGIBILITY:
Inclusion Criteria:

* • Women aged 16 years and older with a good understanding of English

  * Women undergoing a non-emergency elective C/S for a single neonate
  * Pregnancies ≥30 weeks of gestation
  * Taking no regular medication other than pregnancy related vitamins or supplements
  * Participant must be able to give fully informed written consent.

Exclusion Criteria:

* • Significant pregnancy complications or abnormal ultrasound scans

  * Placenta expected to be sent to pathology following delivery (common reasons for this: baby admitted to neonatal unit, abnormal cord blood pH levels, abruption, peripartum sepsis, or severe growth restriction)
  * Any significant disease or disorder in the mother including the following: autoimmune conditions (Lupus, scleroderma, Hashimoto's, RA, arthritis etc), cancer, diabetes, genetic abnormalities, infection (Hepatitis, HIV, EBV, Herpes, STDs, chronic bacterial), liver or kidney disease, neurological conditions or COVID within past 6 months.
  * Currently part of another CTIMP study.
  * Drugs or smoking during pregnancy, or excessive alcohol consumption.
  * Unable to understand English as no translator will be available for this study.
  * Unable to give fully informed consent

Ages: 16 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — All participants must be pregnant biological females and not have undergone gender reassignment
Study Population: Healthy females undergoing a planned C/S for a single neonate (full term)
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-03-08 (Estimated); Primary Completion 2027-07 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Primary outcome measures | From enrolment before Caesarean section to tissue analyses within 12 months
  1. Isolate and grow MSCs from different components of the birth material, such as the chorion, placenta, amniotic fluid, and the umbilical cord.
  2. Collect extracellular vesicles from these different sources of MSCs.
  3. Characterise MSC and EV properties using techniques like microscopy, flow cytometry and ELISAs.
  4. Compare the functions and characteristics of these extracellular vesicles in models of the ageing brain.

CONTACTS AND LOCATIONS:
Locations (1):
- Aberdeen Royal Infirmary, Aberdeen, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
results will be published and can be shared post publication